CLINICAL TRIAL: NCT01101100
Title: A Long-term Assessment of the Safety and Efficacy of AMG 827 Subcutaneous Treatment in Subjects With Psoriasis
Brief Title: Study to Assess the Long-term Safety, Tolerability, and Efficacy of AMG 827 in Subjects With Psoriasis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20090403
Record Dates: First submitted 2010-04-01; First posted 2010-04-09 (Estimated); Results first posted 2019-07-18 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — brodalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AMG 827 (Experimental): AMG 827
  Interventions: Drug: AMG 827

INTERVENTIONS:
Drug: AMG 827 — 210 mg SC or 140 mg SC

SUMMARY:
This study is an open-label extension of study 20090062 to evaluate extended subcutaneous dosing.

DETAILED DESCRIPTION:
This study is an open-label extension of study 20090062 to evaluate extended subcutaneous dosing of AMG 827 for up to 362 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject was randomized into Study 20090062 and completed the week 16 evaluation.

Exclusion Criteria:

* Subject had any Serious Adverse Event (SAE) reported during Study 20090062 that was considered possibly related to IP.
* Subject experienced an adverse event in Study 20090062 that, in the opinion of the investigator, could cause extension of treatment to be detrimental to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2010-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (21):
- United States (6):
  - Research Site, Newnan, Georgia
  - Research Site, Skokie, Illinois
  - Research Site, St Louis, Missouri
  - Research Site, Albuquerque, New Mexico
  - Research Site, Dallas, Texas
  - Research Site, Webster, Texas
- Australia (4):
  - Research Site, Kogarah, New South Wales
  - Research Site, Adelaide, South Australia
  - Research Site, Parkville, Victoria
  - Research Site, Prahran, Victoria
- Canada (6):
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Markham, Ontario
  - Research Site, Waterloo, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Québec, Quebec
- Denmark (2):
  - Research Site, Aarhus
  - Research Site, Hellerup
- France (3):
  - Research Site, Besançon
  - Research Site, Nice
  - Research Site, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Papp K, Leonardi C, Menter A, Thompson EH, Milmont CE, Kricorian G, Nirula A, Klekotka P. Safety and efficacy of brodalumab for psoriasis after 120 weeks of treatment. J Am Acad Dermatol. 2014 Dec;71(6):1183-1190.e3. doi: 10.1016/j.jaad.2014.08.039. Epub 2014 Oct 11. PMID 25313095
- [Derived] Gottlieb A, Lebwohl M, Liu C, Israel RJ, Jacobson A. Malignancy Rates in Brodalumab Clinical Studies for Psoriasis. Am J Clin Dermatol. 2020 Jun;21(3):421-430. doi: 10.1007/s40257-020-00512-4. PMID 32207067
- [Derived] Lebwohl MG, Blauvelt A, Menter A, Papp KA, Guenthner S, Pillai R, Israel RJ, Jacobson A. Efficacy, Safety, and Patient-Reported Outcomes in Patients with Moderate-to-Severe Plaque Psoriasis Treated with Brodalumab for 5 Years in a Long-Term, Open-Label, Phase II Study. Am J Clin Dermatol. 2019 Dec;20(6):863-871. doi: 10.1007/s40257-019-00466-2. PMID 31493163
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label AMG 827: AMG 827: 210 mg SC or 140 mg SC
Period: Overall Study
Arm/Group | Open Label AMG 827
Started | 181
Completed | 126
Not Completed | 55

BASELINE CHARACTERISTICS:
Groups:
- Open Label: AMG 827: 210 mg SC or 140 mg SC
Arm/Group | Open Label
Number analyzed (Participants) | 181
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 173
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 117

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Static Physician's Global Assessment (sPGA) of Clear (0) or Clear/Almost Clear (0 or 1)
Description: Percentage of participants with a static physician's global assessment (sPGA) of clear (0) or clear/almost clear (0 or 1)
Time Frame: 264 weeks
Population: Subjects who were enrolled and had a valid measurement value at the specified week. Results are presented for data up to week 264 as all continuing subjects had completed that visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label AMG 827
Number analyzed (Participants) | 107
Participants | 66

2. Primary Outcome: Percent Change in Psoriasis Area and Severity Index (PASI)
Description: Mean percent change in Psoriasis Area and Severity Index (PASI). A decrease in PASI is an improvement.
Time Frame: 264 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Open Label
Number analyzed (Participants) | 106
Percentage change | -85.7 (26.3)

ADVERSE EVENTS:
Arm/Group | Open Label AMG 827
All-Cause Mortality (participants affected / at risk) | 1/181
Serious Adverse Events (participants affected / at risk) | 29/181
Other Adverse Events (participants affected / at risk) | 177/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label AMG 827 (N=181)
Angina Pectoris (Cardiac disorders) | 1
Myocardial Infaraction (Cardiac disorders) | 3
Hepatitis C (Infections and infestations) | 1
Meningitis Viral (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Duodenal Ulcer (Gastrointestinal disorders) | 1
Pustular Psoriasis (Skin and subcutaneous tissue disorders) | 3
Toxic Skin Eruptions (Skin and subcutaneous tissue disorders) | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1
Cervical Radiculopathy (Nervous system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Abscess (Infections and infestations) | 1
Necrotising fascitis streptococcal (Infections and infestations) | 1
Septic Shock (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastroenteritis eosinophillic (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Intervertabral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Depression (Psychiatric disorders) | 2
Suicidal ideation (Psychiatric disorders) | 1
Aortic aneurysm rupture (Vascular disorders) | 1
Femoral artery occlusion (Vascular disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label AMG 827 (N=181)
Nasopharyngitis (General disorders) | 53
Upper respiratory tract infection (Infections and infestations) | 43
Arthralgia (Musculoskeletal and connective tissue disorders) | 37
Influenza (Infections and infestations) | 28
Back pain (Musculoskeletal and connective tissue disorders) | 26
Gastroenteritis (Gastrointestinal disorders) | 24
Sinusitis (Infections and infestations) | 21
Psoriasis (Skin and subcutaneous tissue disorders) | 19
Hypertension (Nervous system disorders) | 18
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 18
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 18
Muscle strain (Musculoskeletal and connective tissue disorders) | 16
Pain in extremity (General disorders) | 16
Anxiety (Psychiatric disorders) | 15
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 15
Headache (Nervous system disorders) | 14
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 13
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 13
Tendonitis (Musculoskeletal and connective tissue disorders) | 12
Contusion (Injury, poisoning and procedural complications) | 11
Nausea (Gastrointestinal disorders) | 11
Pharyngitis streptococcal (Infections and infestations) | 11
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Fatigue (General disorders) | 10
Insomnia (General disorders) | 10
Nephrolithiasis (Renal and urinary disorders) | 10
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 10
Urinary tract infection (Renal and urinary disorders) | 10
Viral upper respiratory tract infection (Infections and infestations) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other